CLINICAL TRIAL: NCT04330365
Title: Implementation of a Pragmatic Trial of Whole Health Team vs. Primary Care Group Education to Promote Non-Pharmacological Strategies to Improve Pain, Functioning, and Quality of Life in Veterans
Brief Title: Pragmatic Trial of WHT vs. PC-GE to Promote Non-Pharmacological Strategies to Treat Chronic Pain in Veterans
Acronym: wHOPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Francisco Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Karen Seal, Chief of Integrative Medicine, San Francisco Veterans Affairs Medical Center
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: UH3AT009765 (NIH)
Record Dates: First submitted 2020-03-23; First posted 2020-04-01 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Whole Health Team (WHT) Intervention Arm (Active Comparator): The WHT intervention arm includes four core elements: 1) An interdisciplinary WHT collaborating with primary care; 2) Personalized Health Planning with prioritization of multi-modal non-pharmacological and CIH pain management approaches; 3) Whole Health Coaching sessions to assist patients in developing and implementing a Personalized Health Plan for chronic pain care; and 4) the web/mobile Whole Health Resource Directory provided to patient participants (in addition to their providers) to support non-pharmacologic/CIH chronic pain care.
  Interventions: Behavioral: Whole Health Team (WHT) Intervention Arm, Primary Care Group Education (PC-GE) Intervention Arm, Usual Primary Care (UPC) Arm
- Primary Care Group Education (PC-GE) Intervention Arm (Active Comparator): Primary Care Group Education (PC-GE) iss the comparator arm, which is an abbreviated form of Cognitive Behavioral Therapy for Chronic Pain (CBT-CP) adapted for group use in primary care.
  Interventions: Behavioral: Whole Health Team (WHT) Intervention Arm, Primary Care Group Education (PC-GE) Intervention Arm, Usual Primary Care (UPC) Arm
- Usual Primary Care (UPC) Arm (Placebo Comparator): In VA, patient-aligned care teams (PACTs) or primary care is step 1 of VA's Stepped Care Model in the treatment of chronic pain. PCPs are expected to possess the requisite skill set for management of common chronic pain-causing conditions, which includes biopsychosocial assessment, multi-modal treatment, and coordination of specialty pain care after shared-decision making that incorporates patient preferences and values. Participants randomized to this arm will continue to have their PCP and PACT serve in this role.
  Interventions: Behavioral: Whole Health Team (WHT) Intervention Arm, Primary Care Group Education (PC-GE) Intervention Arm, Usual Primary Care (UPC) Arm

INTERVENTIONS:
Behavioral: Whole Health Team (WHT) Intervention Arm, Primary Care Group Education (PC-GE) Intervention Arm, Usual Primary Care (UPC) Arm — Participants will be randomly assigned at the individual level to either WHT, PC-GE or Usual Primary Care, stratified by site, sex, and use of prescribed opioids for chronic pain. The follow-up period for the three arms will be 12 months. The primary outcome is change in pain interference. Secondary outcomes include change in pain intensity, functioning, quality of life, changes in use of pain medications, including opioids (if applicable) and changes in nonpharmacological pain self-management activities. After the baseline assessment, masked telephone assessments will be administered to participants at 3, 6, 9, and 12 months.

SUMMARY:
The overarching goal of this Pain Management Collaboratory Demonstration project is to test a new Whole Health paradigm for chronic pain care, emphasizing non-pharmacological pain self-management that is hypothesized to reduce pain symptoms and improve overall functioning and quality of life in Veterans. In UH3 Aim 1, the investigators will conduct a 12-month pragmatic effectiveness trial at 5 VA sites across the country to test whether veterans with moderate to severe chronic pain randomized to receive the Whole Health Team (WHT) intervention are more likely than those receiving Primary Care Group Education (PC-GE) to: Hypothesis 1: Experience improved pain interference (primary outcome), pain intensity, functioning and quality of life (secondary outcomes); Hypothesis 2: Decrease use of higher-risk pain medications, including opioids, or high-risk combinations; Hypothesis 3: Engage in a greater number of non-pharmacological pain management activities; and Hypothesis 4: Experience improved mental health-related symptoms, including sleep problems and suicidality. In addition, both the WHT and PC-GE arms will be compared to a third group of veterans randomized to Usual Primary Care (UPC, Control) on the same primary and secondary outcomes above. After the baseline assessment, masked telephone assessments will be administered to participants at 3, 6, 9, and 12 months. UH3 Aim 2 is to conduct a process evaluation of the two active interventions (WHT and PC-GE) and a budget impact analysis that includes costs to implement and execute the two active interventions as well as the control condition (UPC) to inform the development of an implementation toolkit for scaling and dissemination. Eligible participants are veterans reporting moderate to severe chronic pain present every day or nearly every day for ≥ 6 months. The total sample size for the population is based on our main study aim/hypothesis and is N=745. This breaks down to n=341 in each of the active interventions (WHT and PC-GE) and N=63 in the Usual Primary Care arm (Control). Results of this UG3/UH3 Pain Management Collaboratory Demonstration project will contribute to the overall mission of the NIH/VA/DoD initiative to build national-level infrastructure that supports non-pharmacologic pain management in veterans and military service personnel.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet the following inclusion criteria to be enrolled in the study:

* Assigned to a VA PCP;
* Report pain present every day or nearly every day for ≥ 6 months using a phone eligibility screener; and
* PEG score of ≥ 5 (including at baseline assessment)

Exclusion Criteria:

Candidates with any of the exclusion criteria at baseline will be excluded from study participation:

* Moderate or severe cognitive impairment as determined by a failed 6-item, validated cognitive screener on initial phone screening (See Appendix A: Telephone Eligibility Screen/Script);
* Active suicidality as determined by medical record review, standardized assessment (PHQ-9) and/or is unable to attend study visits because of an unstable or severe psychiatric or medical condition or is receiving palliative or hospice care; or
* Any other factors that would interfere with study participation including inability to communicate by telephone, VTEL or VVC; being a non-English speaker; plans to relocate within 12 months and concurrent participation in another pain-related study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 793 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2025-01-23 (Actual); Study Completion 2025-01-23 (Actual)

PRIMARY OUTCOMES:
Improved pain interference | 12 months
  The total Brief Pain Inventory (BPI) interference sub-scale score is our primary outcome measure.

SECONDARY OUTCOMES:
Improved pain intensity | 12 months
  Pain intensity rating contained in the 3-item PEG and Brief Pain Inventory (BPI).
Decreased use of higher-risk pain medications, including opioids or high-risk combinations of pain medications (i.e., co-prescription of opioids and benzodiazepines) | 12 months
  The investigators will utilize the VA administrative data/databases to obtain information on prescription medications, including generic name, dispensing information, dose, and instructions.
Engagement in a greater number of non-pharmacological pain management activities | 12 months
  Past-year use of complementary therapies and self-management practices will be measured using the Nonpharmacological and Self-Care Approaches from PMC (NSCAP)185. The inventory assesses use of several CIH modalities such as yoga, etc. The investigators will also probe for other self-directed pain management activities.
Improvement in mental health-related symptoms, including sleep problems and suicidality | 12 months
  The investigators will assess sleep and fatigue symptoms using the PROMIS - Sleep Disturbance. The investigators will be screening for suicidality using the PHQ-9.
Functioning and quality of life | 12 months
  The investigators will assess functioning and quality of life using the THE VETERANS RAND 12-ITEM HEALTH SURVEY (VR-12)

CONTACTS AND LOCATIONS:
Overall Officials: Karen H Seal, MD, Principal Investigator — San Francisco VA Health Care System
Locations (3):
- United States (3):
  - SFVAHCS, San Francisco, California
  - VA St. Louis Health Care System, St Louis, Missouri
  - VAPHCS, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tong G, Seal KH, Becker WC, Li F, Dziura JD, Peduzzi PN, Esserman DA. Impact of complex, partially nested clustering in a three-arm individually randomized group treatment trial: A case study with the wHOPE trial. Clin Trials. 2022 Feb;19(1):3-13. doi: 10.1177/17407745211051288. Epub 2021 Oct 24. PMID 34693748